CLINICAL TRIAL: NCT01438151
Title: Association of Serum Infliximab and Antibodies Toward Infliximab (ATI) to Clinical Outcomes in Crohn's Disease
Brief Title: Understanding the Relationship Between Infliximab Levels to Clinical Response of Remicade in Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated due to poor enrollment
Sponsor: Shradha Agarwal (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Shradha Agarwal, MD, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11-0693
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Remicade; infliximab
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remicade (Experimental): Subjects will begin with receiving infliximab at 5 mg/kg for the first visits. If there is no response to treatment, or flare at any visit (beginning at visit #3), infliximab dose or dosing frequency will be increased in a gradual fashion, up to a maximum of 15 mg/kg every 6 weeks, until response is achieved.
  Interventions: Drug: Remicade

INTERVENTIONS:
Drug: Remicade — The first potential for dose augmentation will be at infusion #3 (visit 1 and 2 patients will receive 5 mg/kg). Patients will be assessed at each infusion visit for response defined as a reduction in HBI score by 2 or more points from prior visit (unless in remission; HBI score of 4 or less). Patients with a response will be maintained at the dose where response was achieved. If there is no response to treatment, or flare at any visit (beginning at visit #3), infliximab dose or dosing frequency will be increased in a gradual fashion, up to a maximum of 15 mg/kg every 6 weeks, until response is achieved.
  Other Names: Dose escalation

SUMMARY:
The purpose of this study is to improve the investigators understanding of the relationship between Crohn's disease and blood levels of the drug infliximab (Remicade). The investigators want to determine whether measuring drug levels can be helpful in understanding how patients respond to this treatment.

DETAILED DESCRIPTION:
The efficacy of infliximab to maintain remission in Crohn's disease has been confirmed by randomized, controlled trials, however the utility of serum infliximab and ATI titers is less clearly described in the clinical practice setting to manage dose and interval levels.

The primary objective of this study is to evaluate the clinical responsiveness of active (HBI >10) Crohn's disease to infliximab as it relates to serum infliximab levels. Though the assay for an infliximab level is commercially available, current dosing practices rely on the assessment of clinical data (laboratory data, symptoms, colonoscopy, etc). In order to understand this relationship, serum infliximab and ATI titers will be collected over the course of 8 (approximately 1 year) infusions. The results of these levels will be retrospectively correlated to the patient's clinical response to treatment.

The secondary objective is to identify predictors of poor response to infliximab by evaluating the efficacy of a dose escalation strategy in patients classified as primary or secondary non-responders.

Understanding the association of serum infliximab levels to disease response may be a useful objective tool to optimize and individualize dosing amount and frequency especially in patients with incomplete or loss of response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active (HBI >10) refractory inflammatory and/or perianal fistulizing Crohn's disease who are prescribed infliximab as standard of care by their gastroenterologist.

Exclusion Criteria:

* Pregnant women.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shradha Agarwal, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Lloyd Mayer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were recruited between 2/16/12 and 10/18/12. Patient were recruited either during inpatient hospitalization or outpatient visit for Remicade.
Groups:
- Remicade: If there is no response to treatment, or flare at any visit (beginning at visit #3), infliximab dose or dosing frequency will be increased in a gradual fashion, up to a maximum of 15 mg/kg every 6 weeks, until response is achieved.
  Remicade: The first potential for dose augmentation will be at infusion #3. Patients will be assessed at each infusion visit for response defined as a reduction in HBI score by 2 or more points from prior visit (unless in remission; HBI score of 4 or less). Patients with a response will be maintained at the dose where response was achieved. If there is no response to treatment, or flare at any visit (beginning at visit #3), infliximab dose or dosing frequency will be increased in a gradual fashion, up to a maximum of 15 mg/kg every 6 weeks, until response is achieved.
Period: Overall Study
Arm/Group | Remicade
Started | 11
Completed | 3
Not Completed | 8
Not completed — study terminated | 8

BASELINE CHARACTERISTICS:
Arm/Group | Remicade
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 34 [10 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Remicade Dose Escalation
Description: At visit 1 and 2, Remicade given at 5mg/kg. If there is no response to treatment, or flare at any visit (beginning at visit #3), infliximab dose or dosing frequency will be increased in a gradual fashion, up to a maximum of 15 mg/kg every 6 weeks, until response is achieved.
Time Frame: 2/16/12-3/22/13
Measure: Number; unit: participants
Arm/Group | Remicade
Number analyzed (Participants) | 11
participants | 5

ADVERSE EVENTS:
Arm/Group | Remicade
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Study was terminated without completion due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days